CLINICAL TRIAL: NCT03200392
Title: The Use Of Er,Cr:YSGG Laser For Recipient Bed Bio-modification And De-epithelialized Palatal Graft Harvesting In The Treatment of Gingival Recession Defects -(Randomized Clinical Trial)
Brief Title: Er,Cr:YSGG Laser For Recipient Bed Bio-modification And Connective Tissue Harvesting in Treatment of Gingival Recession
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Tarek Mahmoud Nasser Eltayeb, laser certified from Aachen University (Germany) and Assistant Lecturer of Periodontology, Oral Medicine and Oral Diagnosis, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 121409
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2017-07

CONDITIONS: Gingival Recession, Localized
Keywords: Er,Cr:YSGG laser; connective tissue graft; root coverage; mucogingival surgery; gingival recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Masking of investigator and participants was not applicable due to surgical procedure and use of laser either for root surface bio-modification or during connective tissue harvesting. The blinded outcome assessor performed the clinical measurements at each selected defect site during the study period. She was not involved in any other part of the study protocol.
Oversight: Data Monitoring Committee: No

ARMS (3):
- L-DGG/LRB (Experimental): laser root surface conditioning & laser DGG harvesting
  Interventions: Device: laser root surface conditioning & laser DGG harvesting
- B-DGG/LRB (Experimental): laser root surface conditioning & blade DGG harvesting
  Interventions: Device: laser root surface conditioning & blade DGG harvesting
- B-DGG (Active Comparator): blade DGG harvesting
  Interventions: Procedure: blade DGG harvesting

INTERVENTIONS:
Device: laser root surface conditioning & laser DGG harvesting — laser root surface bio-modification (single application) and placement of harvested de-epithelialized gingival graft (DGG) followed by coronal repositioned flap for gingival recession Miller's I, II defect coverage
  Other Names: erbium, chromium:YSGG laser
  Arms: L-DGG/LRB
Device: laser root surface conditioning & blade DGG harvesting — laser root surface bio-modification (single application) and scalpel blade harvesting of de-epithelialized palatal graft (Zucchelli et al. 2010) and coronal repositioned flap for gingival recession Miller's I, II defect coverage
  Other Names: erbium, chromium:YSGG laser
  Arms: B-DGG/LRB
Procedure: blade DGG harvesting — De-epithelialized palatal graft harvested using scalpel blade (Zucchelli et al. 2010) and coronal repositioned flap for gingival recession defect coverage
  Arms: B-DGG

SUMMARY:
A clinical and radiographic evaluation of using Erbium, Chromium, Scandium, Gallium and Garnet (Er,Cr:YSGG) laser in recipient site bio-modification and de-epithelialized connective tissue graft harvesting compared to conventional scalpel surgical technique in the treatment of class I and II Miller gingival recession.

DETAILED DESCRIPTION:
Twenty four patients suffering from isolated Class I and II Miller gingival recession defects in anterior esthetic region were enrolled in this study. They were randomly assigned into three groups; de-epithelialized connective tissue graft harvesting technique or; conditioning the exposed root surfaces with Er,Cr:YSGG laser before connective tissue coverage using scalpel blade harvested de-epithelialized connective tissue graft harvesting technique, or; conditioning the exposed root surfaces with the Er,Cr:YSGG laser before Er,Cr:YSGG laser harvested connective tissue using de-epithelialized technique. Clinical and radiographic parameters were recorded at baseline and at 3, 6 and 9 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Single class I, II Miller gingival recession defects (≥ 2mm in depth), presence of identifiable buccal cemento-enamel junction (CEJ) and presence of a step ≤ 1 mm at CEJ.
2. Controlled periodontal disease
3. Full-mouth plaque score of <10%; full-mouth gingival score of <15%
4. Patients available for 9 months follow-up period.

Exclusion Criteria:

1. Smokers.
2. Pregnant and lactating females.
3. Taking medications known to interfere with periodontal tissue health or healing.
4. Previous periodontal surgery on the involved sites.
5. Non-vital teeth.
6. Molar teeth.
7. Recession defects associated with caries or restoration.
8. Occlusal interferences.
9. Taking anti-inflammatory drugs or antibiotics in the past 6 months.

Ages: 21 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in Recession depth | baseline-3-6-9 months
  measured from the gingival margin to the cemento-enamel junction at the mid-buccal aspect of the tooth using William's graduated periodontal probe to the nearest mm

SECONDARY OUTCOMES:
Pain assessment at the donor site | 7 days
  Visual Analogue Scale
number of analgesic pills consumed per day | 7 days
  counting number of analgesic pills per day
Recession width | baseline-3-6-9 months
  distance between mesial and distal gingival margin of the tooth recorded on a horizontal line tangential at the CEJ to the nearest mm
Gingival thickness | baseline and at 9 months
  determined 2mm apical to the gingival margin using standardised CBCT
Height of keratinized tissue width | baseline and at 9 months
  measured form the mid-buccal aspect of the gingival margin to the mucogingival line
Clinical attachment loss | baseline-3-6-9 months
  measured from the CEJ to the bottom of the periodontal pocket to the nearest mm.
Probing pocket depth | baseline-3-6-9 months
  measured from the gingival margin to the base of the periodontal pocket to the nearest mm

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, pHD, Study Chair — Professor Department of Periodontology Ain Shams University; Tarek M Eltayeb, MSc, Principal Investigator — Doctor student Department of Periodontology Misr International University (MIU); Shahinaz G Elashiry, pHD, Study Director — Associate Professor Department of Periodontology MIU; Ramy M Ghali, pHD, Study Director — Professor Department of Prosthodontics Ain Shams University; Fatma H Eldemerdash, pHD, Study Director — Lecturer Department of Periodontology Ain Shams University; Islam S Shaker, MSc, Study Director — Doctor student Department of Oral Radiology MIU
Locations (1):
- Misr International university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ozcelik O, Seydaoglu G, Haytac CM. Diode laser for harvesting de-epithelialized palatal graft in the treatment of gingival recession defects: a randomized clinical trial. J Clin Periodontol. 2016 Jan;43(1):63-71. doi: 10.1111/jcpe.12487. Epub 2016 Jan 21. PMID 26660000